CLINICAL TRIAL: NCT05374265
Title: Cardiovascular Magnetic Resonance Guided Open Artery Trial for Revascularization of Late Presenting ST Elevation Myocardial Infarction: The CRM-OAT Pilot Trial
Brief Title: Cardiovascular Magnetic Resonance Guided Open Artery Trial for Revascularization of Late Presenting ST Elevation Myocardial Infarction
Acronym: CRM-OAT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding Unsuccessful
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STH20171
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Registry (No Intervention): Patients with non-viable myocardium will be treated with standard clinical care.
- OMT with revascularization (Other): Patients with viable myocadium will be randomised to OMT with revascularization. PCI will be performed according to standard techniques using newer generation drug eluting stents. All patients will receive dual anti-platelet treatment for 12 months, or as per local practice guidelines.
  Interventions: Other: Cardiovascular Magnetic Resonance Scan
- OMT alone (Other): Patients with viable myocardium will be radomised to OMT alone. PCI will be performed according to standard techniques using newer generation drug eluting stents. All patients will receive dual anti-platelet treatment for 12 months, or as per local practice guidelines.
  Interventions: Other: Cardiovascular Magnetic Resonance Scan

INTERVENTIONS:
Other: Cardiovascular Magnetic Resonance Scan — Patients will receive a baseline CMR scan to detect viability within 7 days of index admission
  Arms: OMT alone; OMT with revascularization

SUMMARY:
Patients with STEMI are usually treated with primary PCI in contemporary practice. However, primary PCI is currently deemed unbeneficial or potentially harmful in patients presenting late after a STEMI. There is limited data to suggest that patients who may have viable myocardium despite presenting late with a STEMI may derive benefit from PCI, which may be denied in current practice. CMR imaging is the reference modality for assessment of left ventricular function and myocardial viability. This feasibility study will randomise late presenting STEMI patients with CMR documented viability to PCI plus optimal medical therapy (OMT) versus OMT alone. The investigator hypothesises that PCI in this cohort will improve left ventricular remodelling and function. Favourable results will lead to an adequately powered multi-centre trial with the potential to improve the management of late resenting STEMI patients and impact on clinical practice guidelines.

DETAILED DESCRIPTION:
Stable patients with late presenting STEMI will be prospectively recruited into this study from 5 large primary PCI centres in the UK. Ethical approval from a Research Ethics Committee and written informed consent from all participants will be obtained.

Recruited patients will receive baseline CMR to detect viability within 7 days of index admission or coronary angiogram. Patients with non-viable myocardium will be treated with standard clinical care and form part of the registry arm. Patients with viable myocardium will be randomised to revascularization with OMT vs OMT alone. PCI will be performed according to standard techniques using newer generation drug eluting stents. All patients will recieve dual anti-platelet treatment for 12 months, or as per local practice guidelines. other treatments will be given according to evidence based guidelines. Revascularization wth CABG can also be considered, based on MDT decision.

The feasibility study will randomise 60 patients (30 in PCI and 30 in OMT group). OAT-NUC trial showed that 70% late presenting STEMI may have viability. therefor, recruiting 90 patients for baseline CMR may provide 60 patients to randomise. the results of this feasibility study will inform the investigator of the numbers needed for an adequately powered multi-centre clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients presenting >12 hours, and within 28 days, after symptom onsent.
* Stable patients with no on-going features of ischaemia (chest pain, dynamic ECG changes)

Exclusion Criteria:

* Inability to give informed consent
* Standard CMR contra-indications
* Haemodynamic instability (requiring on-going intravenous therapy or respiratory support)
* Previous coronary artery bypass grafting and cardiomyopathy
* Estimated glomerular filtration rate <30ml/min/1.73m2
* End-stage malignancy or expected life expectancy of less than 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in LV end-systolic volume | from baseline to 3-months
  Change in LV end-systolic volume from baseline to 3-month CMR.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Hospitals NHS FT, Sheffield, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Background] O'Gara PT, Kushner FG, Ascheim DD, Casey DE Jr, Chung MK, de Lemos JA, Ettinger SM, Fang JC, Fesmire FM, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX. 2013 ACCF/AHA guideline for the management of ST-elevation myocardial infarction: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Jan 29;61(4):e78-e140. doi: 10.1016/j.jacc.2012.11.019. Epub 2012 Dec 17. No abstract available. PMID 23256914
- [Background] Eagle KA, Goodman SG, Avezum A, Budaj A, Sullivan CM, Lopez-Sendon J; GRACE Investigators. Practice variation and missed opportunities for reperfusion in ST-segment-elevation myocardial infarction: findings from the Global Registry of Acute Coronary Events (GRACE). Lancet. 2002 Feb 2;359(9304):373-7. doi: 10.1016/S0140-6736(02)07595-5. PMID 11844506
- [Background] Schiele F, Hochadel M, Tubaro M, Meneveau N, Wojakowski W, Gierlotka M, Polonski L, Bassand JP, Fox KA, Gitt AK. Reperfusion strategy in Europe: temporal trends in performance measures for reperfusion therapy in ST-elevation myocardial infarction. Eur Heart J. 2010 Nov;31(21):2614-24. doi: 10.1093/eurheartj/ehq305. Epub 2010 Aug 30. PMID 20805111
- [Background] Dzavik V, Beanlands DS, Davies RF, Leddy D, Marquis JF, Teo KK, Ruddy TD, Burton JR, Humen DP. Effects of late percutaneous transluminal coronary angioplasty of an occluded infarct-related coronary artery on left ventricular function in patients with a recent (< 6 weeks) Q-wave acute myocardial infarction (Total Occlusion Post-Myocardial Infarction Intervention Study [TOMIIS]--a pilot study). Am J Cardiol. 1994 May 1;73(12):856-61. doi: 10.1016/0002-9149(94)90809-5. PMID 8184807
- [Background] Horie H, Takahashi M, Minai K, Izumi M, Takaoka A, Nozawa M, Yokohama H, Fujita T, Sakamoto T, Kito O, Okamura H, Kinoshita M. Long-term beneficial effect of late reperfusion for acute anterior myocardial infarction with percutaneous transluminal coronary angioplasty. Circulation. 1998 Dec 1;98(22):2377-82. doi: 10.1161/01.cir.98.22.2377. PMID 9832481
- [Background] Silva JC, Rochitte CE, Junior JS, Tsutsui J, Andrade J, Martinez EE, Moffa PJ, Menegheti JC, Kalil-Filho R, Ramires JF, Nicolau JC. Late coronary artery recanalization effects on left ventricular remodelling and contractility by magnetic resonance imaging. Eur Heart J. 2005 Jan;26(1):36-43. doi: 10.1093/eurheartj/ehi011. Epub 2004 Nov 29. PMID 15615797
- [Background] Yousef ZR, Redwood SR, Bucknall CA, Sulke AN, Marber MS. Late intervention after anterior myocardial infarction: effects on left ventricular size, function, quality of life, and exercise tolerance: results of the Open Artery Trial (TOAT Study). J Am Coll Cardiol. 2002 Sep 4;40(5):869-76. doi: 10.1016/s0735-1097(02)02058-2. PMID 12225709
- [Background] Steg PG, Thuaire C, Himbert D, Carrie D, Champagne S, Coisne D, Khalife K, Cazaux P, Logeart D, Slama M, Spaulding C, Cohen A, Tirouvanziam A, Montely JM, Rodriguez RM, Garbarz E, Wijns W, Durand-Zaleski I, Porcher R, Brucker L, Chevret S, Chastang C; DECOPI Investigators. DECOPI (DEsobstruction COronaire en Post-Infarctus): a randomized multi-centre trial of occluded artery angioplasty after acute myocardial infarction. Eur Heart J. 2004 Dec;25(24):2187-94. doi: 10.1016/j.ehj.2004.10.019. PMID 15589635
- [Background] Hochman JS, Lamas GA, Buller CE, Dzavik V, Reynolds HR, Abramsky SJ, Forman S, Ruzyllo W, Maggioni AP, White H, Sadowski Z, Carvalho AC, Rankin JM, Renkin JP, Steg PG, Mascette AM, Sopko G, Pfisterer ME, Leor J, Fridrich V, Mark DB, Knatterud GL; Occluded Artery Trial Investigators. Coronary intervention for persistent occlusion after myocardial infarction. N Engl J Med. 2006 Dec 7;355(23):2395-407. doi: 10.1056/NEJMoa066139. Epub 2006 Nov 14. PMID 17105759
- [Background] Hochman JS, Reynolds HR, Dzavik V, Buller CE, Ruzyllo W, Sadowski ZP, Maggioni AP, Carvalho AC, Rankin JM, White HD, Goldberg S, Forman SA, Mark DB, Lamas GA; Occluded Artery Trial Investigators. Long-term effects of percutaneous coronary intervention of the totally occluded infarct-related artery in the subacute phase after myocardial infarction. Circulation. 2011 Nov 22;124(21):2320-8. doi: 10.1161/CIRCULATIONAHA.111.041749. Epub 2011 Oct 24. PMID 22025606
- [Background] Dzavik V, Buller CE, Lamas GA, Rankin JM, Mancini GB, Cantor WJ, Carere RJ, Ross JR, Atchison D, Forman S, Thomas B, Buszman P, Vozzi C, Glanz A, Cohen EA, Meciar P, Devlin G, Mascette A, Sopko G, Knatterud GL, Hochman JS; TOSCA-2 Investigators. Randomized trial of percutaneous coronary intervention for subacute infarct-related coronary artery occlusion to achieve long-term patency and improve ventricular function: the Total Occlusion Study of Canada (TOSCA)-2 trial. Circulation. 2006 Dec 5;114(23):2449-57. doi: 10.1161/CIRCULATIONAHA.106.669432. Epub 2006 Nov 14. PMID 17105848
- [Background] Ioannidis JP, Katritsis DG. Percutaneous coronary intervention for late reperfusion after myocardial infarction in stable patients. Am Heart J. 2007 Dec;154(6):1065-71. doi: 10.1016/j.ahj.2007.07.049. Epub 2007 Sep 14. PMID 18035076
- [Background] Udelson JE, Pearte CA, Kimmelstiel CD, Kruk M, Kufera JA, Forman SA, Teresinska A, Bychowiec B, Marin-Neto JA, Hochtl T, Cohen EA, Caramori P, Busz-Papiez B, Adlbrecht C, Sadowski ZP, Ruzyllo W, Kinan DJ, Lamas GA, Hochman JS. The Occluded Artery Trial (OAT) Viability Ancillary Study (OAT-NUC): influence of infarct zone viability on left ventricular remodeling after percutaneous coronary intervention versus optimal medical therapy alone. Am Heart J. 2011 Mar;161(3):611-21. doi: 10.1016/j.ahj.2010.11.020. PMID 21392619
- [Background] Ibrahim T, Bulow HP, Hackl T, Hornke M, Nekolla SG, Breuer M, Schomig A, Schwaiger M. Diagnostic value of contrast-enhanced magnetic resonance imaging and single-photon emission computed tomography for detection of myocardial necrosis early after acute myocardial infarction. J Am Coll Cardiol. 2007 Jan 16;49(2):208-16. doi: 10.1016/j.jacc.2006.08.047. Epub 2006 Dec 29. PMID 17222732
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Bellenger NG, Yousef Z, Rajappan K, Marber MS, Pennell DJ. Infarct zone viability influences ventricular remodelling after late recanalisation of an occluded infarct related artery. Heart. 2005 Apr;91(4):478-83. doi: 10.1136/hrt.2004.034918. PMID 15772205
- [Background] Malek LA, Silva JC, Bellenger NG, Nicolau JC, Klopotowski M, Spiewak M, Rassi CH, Lewandowski Z, Kruk M, Rochitte CE, Ruzyllo W, Witkowski A. Late percutaneous coronary intervention for an occluded infarct-related artery in patients with preserved infarct zone viability: a pooled analysis of cardiovascular magnetic resonance studies. Cardiol J. 2013;20(5):552-9. doi: 10.5603/CJ.2013.0141. PMID 24297771
- [Background] Deyell MW, Buller CE, Miller LH, Wang TY, Dai D, Lamas GA, Srinivas VS, Hochman JS. Impact of National Clinical Guideline recommendations for revascularization of persistently occluded infarct-related arteries on clinical practice in the United States. Arch Intern Med. 2011 Oct 10;171(18):1636-43. doi: 10.1001/archinternmed.2011.315. Epub 2011 Jul 11. PMID 21747002
- [Background] Bodi V, Sanchis J, Nunez J, Mainar L, Lopez-Lereu MP, Monmeneu JV, Rumiz E, Chaustre F, Trapero I, Husser O, Forteza MJ, Chorro FJ, Llacer A. Prognostic value of a comprehensive cardiac magnetic resonance assessment soon after a first ST-segment elevation myocardial infarction. JACC Cardiovasc Imaging. 2009 Jul;2(7):835-42. doi: 10.1016/j.jcmg.2009.03.011. PMID 19608133
- [Background] Kim RJ, Fieno DS, Parrish TB, Harris K, Chen EL, Simonetti O, Bundy J, Finn JP, Klocke FJ, Judd RM. Relationship of MRI delayed contrast enhancement to irreversible injury, infarct age, and contractile function. Circulation. 1999 Nov 9;100(19):1992-2002. doi: 10.1161/01.cir.100.19.1992. PMID 10556226
- [Background] Kim RJ, Wu E, Rafael A, Chen EL, Parker MA, Simonetti O, Klocke FJ, Bonow RO, Judd RM. The use of contrast-enhanced magnetic resonance imaging to identify reversible myocardial dysfunction. N Engl J Med. 2000 Nov 16;343(20):1445-53. doi: 10.1056/NEJM200011163432003. PMID 11078769
- [Background] Choi KM, Kim RJ, Gubernikoff G, Vargas JD, Parker M, Judd RM. Transmural extent of acute myocardial infarction predicts long-term improvement in contractile function. Circulation. 2001 Sep 4;104(10):1101-7. doi: 10.1161/hc3501.096798. PMID 11535563
- [Background] Ugander M, Bagi PS, Oki AJ, Chen B, Hsu LY, Aletras AH, Shah S, Greiser A, Kellman P, Arai AE. Myocardial edema as detected by pre-contrast T1 and T2 CMR delineates area at risk associated with acute myocardial infarction. JACC Cardiovasc Imaging. 2012 Jun;5(6):596-603. doi: 10.1016/j.jcmg.2012.01.016. PMID 22698528
- [Background] Bulluck H, White SK, Rosmini S, Bhuva A, Treibel TA, Fontana M, Abdel-Gadir A, Herrey A, Manisty C, Wan SM, Groves A, Menezes L, Moon JC, Hausenloy DJ. T1 mapping and T2 mapping at 3T for quantifying the area-at-risk in reperfused STEMI patients. J Cardiovasc Magn Reson. 2015 Aug 12;17(1):73. doi: 10.1186/s12968-015-0173-6. PMID 26264813
- [Background] Stork A, Lund GK, Muellerleile K, Bansmann PM, Nolte-Ernsting C, Kemper J, Begemann PG, Adam G. Characterization of the peri-infarction zone using T2-weighted MRI and delayed-enhancement MRI in patients with acute myocardial infarction. Eur Radiol. 2006 Oct;16(10):2350-7. doi: 10.1007/s00330-006-0232-3. Epub 2006 Apr 20. PMID 16625349
- [Background] Kidambi A, Motwani M, Uddin A, Ripley DP, McDiarmid AK, Swoboda PP, Broadbent DA, Musa TA, Erhayiem B, Leader J, Croisille P, Clarysse P, Greenwood JP, Plein S. Myocardial Extracellular Volume Estimation by CMR Predicts Functional Recovery Following Acute MI. JACC Cardiovasc Imaging. 2017 Sep;10(9):989-999. doi: 10.1016/j.jcmg.2016.06.015. Epub 2016 Oct 19. PMID 27771398
- [Background] Bulluck H, Rosmini S, Abdel-Gadir A, Bhuva AN, Treibel TA, Fontana M, Knight DS, Nordin S, Sirker A, Herrey AS, Manisty C, Moon JC, Hausenloy DJ. Redefining viability by cardiovascular magnetic resonance in acute ST-segment elevation myocardial infarction. Sci Rep. 2017 Nov 7;7(1):14676. doi: 10.1038/s41598-017-15353-1. PMID 29116176